CLINICAL TRIAL: NCT03475108
Title: Integrating Community Health Workers Into the Care of Children With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-014828
Record Dates: First submitted 2018-03-12; First posted 2018-03-23 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes Mellitus; Psychosocial Problem; Compliance, Patient; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Patient Compliance; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Crossover Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Health Worker Group (Experimental): Patients are assigned a community health worker for one year, in addition to standard diabetes care. They do not receive a community health worker for the second year of the study.
  Interventions: Other: Community Health Worker added to diabetes team
- Standard Diabetes Care Group (Other): Patients receive standard diabetes care for one year. They receive a community health worker for the second year (as part of a crossover trial).
  Interventions: Other: Community Health Worker added to diabetes team

INTERVENTIONS:
Other: Community Health Worker added to diabetes team — A Community Health Worker will be added to the diabetes team caring for a child with type 1 diabetes over 1 year. The intervention includes social determinants of health screening and goal setting, with home visits.

SUMMARY:
The primary aim of this randomized controlled trial is to determine if the integration of a Community Health Worker into the healthcare team is associated with an improvement in diabetes control in children with type 1 diabetes. The secondary objectives are to determine if utilization of Community Health Workers is also associated with reduced emergency department visits and hospitalizations, improved attendance at outpatient diabetes appointments, and improvements in psychosocial outcomes and diabetes control.

DETAILED DESCRIPTION:
Diabetic ketoacidosis accounts for 65% of hospitalizations in pediatric patients with type 1 diabetes, and has a mortality rate between 0.15-0.31%. Children with established type 1 diabetes have an 8% annualized risk of developing diabetic ketoacidosis, and this risk increases during adolescence. In addition, socioeconomic and racial disparities are associated with increased risks of poor glycemic control, hospitalization with diabetic ketoacidosis, and even severe hypoglycemia. All of these complications are associated with preventable harm, and lead to increased utilization of medical resources, both in the short- and long-term. Social determinants of health account for over 75% of health outcomes. Thus, it is not surprising that a disproportionate number of children with poor diabetes control and recurrent hospitalization in diabetic ketoacidosis come from vulnerable underserved populations.

In this study, Investigators will study the effect of integrating a community-based healthcare worker into the healthcare team of children with poorly controlled type 1 diabetes. Community Health Workers (CHW) are highly motivated, community members who do not necessarily have prior medical training, but rather they link with the healthcare team to identify and provide relevant social supports to the family. They receive specific training that focuses on issues relevant to improving health outcomes and adherence, by improving medication access, reducing food insecurity, and improving health literacy. The CHW are able to provide real-time assistance with navigating the healthcare and social services systems, reducing family stress and breaking down community barriers to positive health behavior. The CHW work with the family to develop goals and develop an individualized plan to reach these goals. The role of the CHW can include home visits, phone contacts, meeting with school representatives and accompanying patients to appointments.

At the diabetes center at The Children's Hospital of Philadelphia (CHOP), the Community Health Worker will be assigned for one year to patients with high healthcare utilization and / or poorly controlled type 1 diabetes. The support provided for this year will be tailored to the patient's needs but may include problem solving surrounding issues related to work/education, accessing healthcare/medications, engagement with the healthcare team, transportation, housing or food insecurity. Interactions with patients will be through home visits, telephone encounters, text messaging or email. This will be added to their medical care and will be documented in the patient's medical record.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of type 1 diabetes for > 1 year
* Either:

Over the previous one year, the sum of the following should be > 2: diabetes-related hospitalizations plus emergency department visits plus missed appointments (on separate days) or Hemoglobin A1c ≥ 9.5 at the time of enrollment.

Exclusion Criteria:

* Children in custody of the State where there is no identified caretaker who can complete study procedures

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 2 years
  Improvement in glycemic control, as measured by hemoglobin A1c

SECONDARY OUTCOMES:
Hospital admissions | 2 years
  Data will be extracted from the medical record of each patient to obtain information on the number of hospital admissions.
Attended outpatient appointments | 2 years
  Data will be extracted from the medical record of each patient to obtain information on the number of attended outpatient appointments.
Missed outpatient appointments | 2 years
  Data will be extracted from the medical record of each patient to obtain information on the number of missed outpatient appointments.
Emergency Department utilization | 2 years
  Data will be extracted from the medical record of each patient to obtain information about the number of Emergency Department (ED) visits.
Primary caregiver's diabetes self-efficacy | 2 years
  The 17-item, "Parental self efficacy in diabetes scale" will be completed by the primary caregiver using a 5-point Likert rating scale. The questionnaire will provide information to assess glycemic control, and sub analysis of results related to diabetes management, problem solving and teaching. This scale ranges in score from 17 to 85, with higher scores consistent with increased self-efficacy.
Quality of life (primary care giver) | 2 years
  The primary care giver will complete the 36-item "PedsQL Health related quality of life for parents of children with chronic disease" questionnaire (HCCQ) using a 5-point Likert rating scale to assess how their child's illness has had an impact on their quality of life. This scale ranges in score from 0 to 144, with higher scores consistent with decreased quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Colin P Hawkes, MD PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rewers A, Chase HP, Mackenzie T, Walravens P, Roback M, Rewers M, Hamman RF, Klingensmith G. Predictors of acute complications in children with type 1 diabetes. JAMA. 2002 May 15;287(19):2511-8. doi: 10.1001/jama.287.19.2511. PMID 12020331
- [Background] Hassan K, Loar R, Anderson BJ, Heptulla RA. The role of socioeconomic status, depression, quality of life, and glycemic control in type 1 diabetes mellitus. J Pediatr. 2006 Oct;149(4):526-31. doi: 10.1016/j.jpeds.2006.05.039. PMID 17011326
- [Background] Kangovi S, Mitra N, Grande D, White ML, McCollum S, Sellman J, Shannon RP, Long JA. Patient-centered community health worker intervention to improve posthospital outcomes: a randomized clinical trial. JAMA Intern Med. 2014 Apr;174(4):535-43. doi: 10.1001/jamainternmed.2013.14327. PMID 24515422
- [Background] Laffel LM, Brackett J, Ho J, Anderson BJ. Changing the process of diabetes care improves metabolic outcomes and reduces hospitalizations. Qual Manag Health Care. 1998 Sep;6(4):53-62. doi: 10.1097/00019514-199806040-00006. PMID 10339045
- [Background] Raphael JL, Rueda A, Lion KC, Giordano TP. The role of lay health workers in pediatric chronic disease: a systematic review. Acad Pediatr. 2013 Sep-Oct;13(5):408-20. doi: 10.1016/j.acap.2013.04.015. PMID 24011745